CLINICAL TRIAL: NCT01803555
Title: A 12-Week Efficacy and Safety Evaluation of Budesonide/Formoterol SPIROMAX(R) 160/4.5 mcg Inhalation Powder Versus SYMBICORT(R) TURBOHALER(R) 200/6 mcg in Adult and Adolescent Patients With Persistent Asthma
Brief Title: Efficacy and Safety Evaluation of Budesonide/Formoterol SPIROMAX® Inhalation Powder Versus SYMBICORT® TURBOHALER®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BFS-AS-306
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Results first posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-03

CONDITIONS: Asthma
Keywords: Budesonide/Formoterol SPIROMAX®; SYMBICORT® TURBOHALER®; Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BF Spiromax (Experimental): 2 inhalations of BF Spiromax at a dosage of 160/4.5 mcg and 2 inhalations of SYMBICORT placebo administered twice daily (AM and PM) during the 12-week treatment period.
  Interventions: Drug: Budesonide/Formoterol SPIROMAX®; Drug: SYMBICORT placebo
- Symbicort Turbohaler (Active Comparator): 2 inhalations of SYMBICORT TURBOHALER at a dosage of 200/6 mcg and 2 inhalations of placebo SPIROMAX administered twice daily (AM and PM) during the 12-week treatment period.
  Interventions: Drug: SYMBICORT® TURBOHALER®; Drug: SPIROMAX Placebo

INTERVENTIONS:
Drug: Budesonide/Formoterol SPIROMAX® — BF Spiromax will be administered per dose and schedule specified in the arm.
  Arms: BF Spiromax
Drug: SYMBICORT® TURBOHALER® — Symbicort Turbohaler will be administered per dose and schedule specified in the arm.
  Arms: Symbicort Turbohaler
Drug: SYMBICORT placebo — SYMBICORT placebo multi-dose dry powder inhaler (DPI) identical in appearance to SYMBICORT TURBOHALER will be administered per dose and schedule specified in the arm.
  Arms: BF Spiromax
Drug: SPIROMAX Placebo — SPIROMAX Placebo multi-dose dry powder inhaler (DPI) identical in appearance to BF SPIROMAX will be administered per dose and schedule specified in the arm.
  Arms: Symbicort Turbohaler

SUMMARY:
The primary objective of the study is to establish whether budesonide/formoterol fumarate dihydrate (BF) Spiromax 160/4.5 micrograms (mcg) is as effective as Symbicort Turbohaler 200/6 mcg administered twice daily in participants with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 12 years and older as of the screening visit. Male or female participants 18 years and older, as of the screening visit, in countries where local regulations or the regulatory status of study medication permit enrollment of adult participants only.
* General good health, and free of any concomitant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the participant at increased risk during the study.
* Asthma Diagnosis: The asthma diagnosis must be in accordance with the Global Initiative for Asthma (GINA)

Exclusion Criteria:

* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures.
* Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear that is not resolved within 2 weeks before the screening visit. In addition, the participant must be excluded if such infection occurs between the screening visit and the baseline visit.
* Any asthma exacerbation requiring oral corticosteroids within 1 month of the screening visit. A participant must not have been hospitalized for asthma within 6 months before the screening visit.
* Presence of glaucoma, cataracts, ocular herpes simplex, or malignancy other than basal cell carcinoma.
* Historical or current evidence of a clinically significant disease including, but not limited to: cardiovascular conditions (for example, congestive heart failure, known aortic aneurysm, clinically significant cardiac arrhythmia or coronary heart disease), hepatic, renal, hematological, neuropsychological, endocrine conditions (for example, uncontrolled diabetes mellitus, uncontrolled thyroid disorder, Addison's disease, Cushing's syndrome), gastrointestinal conditions (for example, poorly-controlled peptic ulcer, gastroesophageal reflux disease [GERD]), or pulmonary conditions (for example, chronic bronchitis, emphysema, bronchiectasis with the need for treatment, cystic fibrosis, bronchopulmonary dysplasia, chronic obstructive pulmonary disease). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the participant at risk through participation, or which could affect the efficacy or safety analysis if the disease/condition became exacerbated during the study.

NOTE: Other inclusion and exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2013-07-04 (Actual); Primary Completion 2014-03-20 (Actual); Study Completion 2014-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, M.D., Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (114):
- Austria (3):
  - Teva Investigational Site 33020, Grieskirchen
  - Teva Investigational Site 33019, Linz
  - Teva Investigational Site 33018, Wels
- Belgium (3):
  - Teva Investigational Site 37029, Gozée
  - Teva Investigational Site 37031, Halen
  - Teva Investigational Site 37030, Jambes
- Czechia (9):
  - Teva Investigational Site 54056, Brno
  - Teva Investigational Site 54061, Hradec Králové
  - Teva Investigational Site 54068, Neratovice
  - Teva Investigational Site 54063, Ostrava - Marianske Hory
  - Teva Investigational Site 54065, Pilsen
  - Teva Investigational Site 54067, Prague
  - Teva Investigational Site 54058, Prague
  - Teva Investigational Site 54064, Rokycany
  - Teva Investigational Site 54059, Strakonice
- Denmark (2):
  - Teva Investigational Site 39020, Copenhagen NV
  - Teva Investigational Site 39021, Odense
- Finland (5):
  - Teva Investigational Site 40004, Helsinki
  - Teva Investigational Site 40005, Jyväskylä
  - Teva Investigational Site 40002, Pori
  - Teva Investigational Site 40001, Tampere
  - Teva Investigational Site 40003, Turku
- France (6):
  - Teva Investigational Site 35088, Brest
  - Teva Investigational Site 35089, La Bouëxière
  - Teva Investigational Site 35093, Lyon
  - Teva Investigational Site 35092, Mûrs-Erigné
  - Teva Investigational Site 35090, Nantes
  - Teva Investigational Site 35091, Perpignan
- Germany (17):
  - Teva Investigational Site 32243, Berlin
  - Teva Investigational Site 32255, Berlin
  - Teva Investigational Site 32256, Berlin
  - Teva Investigational Site 32257, Berlin
  - Teva Investigational Site 32252, Cottbus
  - Teva Investigational Site 32251, Frankfurt am Main
  - Teva Investigational Site 32253, Frankfurt am Main
  - Teva Investigational Site 32254, Gelsenkirchen
  - Teva Investigational Site 32259, Großhansdorf
  - Teva Investigational Site 32249, Hamburg
  - Teva Investigational Site 32246, Leipzig
  - Teva Investigational Site 32240, Neu-Isenburg
  - Teva Investigational Site 32244, Neukölln
  - Teva Investigational Site 32258, Offenbach
  - Teva Investigational Site 32250, Reinfeld
  - Teva Investigational Site 32241, Rüdersdorf
  - Teva Investigational Site 32247, Weinheim
- Hungary (11):
  - Teva Investigational Site 51075, Balassagyarmat
  - Teva Investigational Site 51072, Budapest
  - Teva Investigational Site 51067, Budapest
  - Teva Investigational Site 51077, Csorna
  - Teva Investigational Site 51065, Deszk
  - Teva Investigational Site 51071, Kaposvár
  - Teva Investigational Site 51073, Kaposvár
  - Teva Investigational Site 51068, Komárom
  - Teva Investigational Site 51070, Mosdós
  - Teva Investigational Site 51076, Tatabánya
  - Teva Investigational Site 51074, Törökbálint
- Israel (7):
  - Teva Investigational Site 80036, Afula
  - Teva Investigational Site 80035, Haifa
  - Teva Investigational Site 80040, Kfar Saba
  - Teva Investigational Site 80039, Petah Tikva
  - Teva Investigational Site 80037, Ramat Gan
  - Teva Investigational Site 80038, Rehovot
  - Teva Investigational Site 80041, Ẕerifin
- Italy (3):
  - Teva Investigational Site 30055, Cisanello Pisa
  - Teva Investigational Site 30056, Milan
  - Teva Investigational Site 30054, Padua
- Netherlands (2):
  - Teva Investigational Site 38048, Alkmaar
  - Teva Investigational Site 38049, Leeuwarden
- Poland (19):
  - Teva Investigational Site 53114, Bialystok
  - Teva Investigational Site 53110, Bialystok
  - Teva Investigational Site 53117, Gdansk
  - Teva Investigational Site 53106, Gdansk
  - Teva Investigational Site 53109, Krakow
  - Teva Investigational Site 53111, Krakow
  - Teva Investigational Site 53100, Krakow
  - Teva Investigational Site 53107, Lodz
  - Teva Investigational Site 53102, Lublin
  - Teva Investigational Site 53116, Poznan
  - Teva Investigational Site 53119, Sopot
  - Teva Investigational Site 53103, Strzelce Opolskie
  - Teva Investigational Site 53104, Szczecin
  - Teva Investigational Site 53105, Tarnów
  - Teva Investigational Site 53120, Wroclaw
  - Teva Investigational Site 53099, Wroclaw
  - Teva Investigational Site 53115, Wroclaw
  - Teva Investigational Site 53113, Zabrze
  - Teva Investigational Site 53101, Zgierz
- Russia (9):
  - Teva Investigational Site 50179, Kazan'
  - Teva Investigational Site 50177, Moscow
  - Teva Investigational Site 50178, Saint Petersburg
  - Teva Investigational Site 50175, Saint Petersburg
  - Teva Investigational Site 50171, Saint Petersburg
  - Teva Investigational Site 50172, Saratov
  - Teva Investigational Site 50173, Tomsk
  - Teva Investigational Site 50170, Vsevolozhsk
  - Teva Investigational Site 50174, Yaroslavl
- Spain (9):
  - Teva Investigational Site 31051, Alcorcón
  - Teva Investigational Site 31054, Badalona
  - Teva Investigational Site 31052, Barcelona
  - Teva Investigational Site 31057, Barcelona
  - Teva Investigational Site 31053, Bilbao
  - Teva Investigational Site 31058, Madrid
  - Teva Investigational Site 31056, Pamplona
  - Teva Investigational Site 31055, Seville
  - Teva Investigational Site 31061, Vitoria-Gasteiz
- Sweden (3):
  - Teva Investigational Site 42014, Gothenburg
  - Teva Investigational Site 42011, Lund
  - Teva Investigational Site 42012, Stockholm
- United Kingdom (6):
  - Teva Investigational Site 34024, Chesterfield
  - Teva Investigational Site 34026, Coventry
  - Teva Investigational Site 34022, Dundee
  - Teva Investigational Site 34027, East Sussex
  - Teva Investigational Site 34029, Lancashire
  - Teva Investigational Site 34028, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.

REFERENCES:
- [Derived] Virchow JC, Rodriguez-Roisin R, Papi A, Shah TP, Gopalan G. A randomized, double-blinded, double-dummy efficacy and safety study of budesonide-formoterol Spiromax(R) compared to budesonide-formoterol Turbuhaler(R) in adults and adolescents with persistent asthma. BMC Pulm Med. 2016 Mar 17;16:42. doi: 10.1186/s12890-016-0200-x. PMID 26987997

RESULTS

PARTICIPANT FLOW:
Groups:
- BF Spiromax: Participants received budesonide/formoterol Spiromax (BF)(budesonide/formoterol fumarate dihydrate 160/4.5 micrograms [mcg]) 2 inhalations twice daily and Symbicort placebo 2 inhalations twice daily for 12 weeks.
- Symbicort Turbohaler: Participants received Symbicort Turbohaler (budesonide/formoterol fumarate dihydrate 200/6 mcg) 2 inhalations twice daily and placebo Spiromax 2 inhalations twice daily for 12 weeks.
Period: Overall Study
Arm/Group | BF Spiromax | Symbicort Turbohaler
Started | 303 | 302
Received at Least 1 Dose of Study Drug | 303 | 299
Completed | 290 | 284
Not Completed | 13 | 18
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Non-compliance | 1 | 1
Not completed — Protocol Violation | 3 | 5
Not completed — Lost to Follow-up | 0 | 2
Not completed — Other than specified | 3 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | BF Spiromax | Symbicort Turbohaler | Total
Number analyzed (Participants) | 303 | 302 | 605
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (16.24) | 46.9 (16.89) | 47.5 (16.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 161 | 333
  Male | 131 | 141 | 272
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 297 | 299 | 596
  Unknown or Not Reported | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 297 | 300 | 597
  Black | 2 | 1 | 3
  Asian | 1 | 1 | 2
  American Indian or Alaskan Native | 0 | 0 | 0
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Other | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weekly Average of Daily Trough (Predose and Pre-rescue Bronchodilator) Morning (AM) Peak Expiratory Flow (PEF) Over the 12-Week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Baseline trough morning PEF was defined as the average value of recorded (nonmissing) morning assessments 5 out of the last 7 days prior to randomization. The first day before randomization consisted of the electronic patient diary entry at home on the morning of the randomization visit (Baseline [Day 1]) and the first day postrandomization consisted of the electronic patient diary entry at home on the morning of the day after the randomization visit (Baseline [Day 1]). For postdose weekly average of trough morning PEF measurements, the values were the averages based on the available data for that week. The averages were calculated as the sum of morning PEF values divided by the number of nonmissing assessments. The final value for change from baseline was calculated as the average of the weekly change from baseline averaged over 12 weeks.
Time Frame: Baseline, Weeks 1 to 12 (averaged over 12 weeks)
Population: The per-protocol (PP) population included all data from randomized participants obtained before experiencing major protocol deviations (that is, protocol violations). Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: liters (L)/minute (min)
Arm/Group | BF Spiromax | Symbicort Turbohaler
Number analyzed (Participants) | 289 | 284
liters (L)/minute (min) | 18.839 (2.754) | 21.796 (2.745)
Statistical Analysis 1: Comparison: BF Spiromax vs Symbicort Turbohaler; Test type: Non-Inferiority — The noninferiority of BF Spiromax to Symbicort Turbohaler was demonstrated if the lower limit of the 2-sided 95% confidence interval (CI) for the treatment difference was greater than -15 L/min; p = 0.3387, Mixed Models Analysis; Analysis included effects due to baseline weekly average of daily trough AM PEF, gender, age, treatment, time, and treatment-by-time interaction; Least Square (LS) mean difference = -2.957, 95% CI 2-sided [-9.02 to 3.11]

2. Secondary Outcome: Change From Baseline in Weekly Average of Daily Evening (PM) PEF Over the 12-Week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. Baseline was defined as the average value of the recorded (nonmissing) assessments over the 7 days prior to randomization. For postdose weekly average of evening PEF measurements, the values were the averages based on the available data for that week. The averages were calculated as the sum of evening PEF values divided by the number of nonmissing assessments. The final value for change from baseline was calculated as the average of the weekly change from baseline averaged over 12 weeks.
Time Frame: Baseline, Weeks 1 to 12 (averaged over 12 weeks)
Population: The PP population included all data from randomized participants obtained before experiencing major protocol deviations (that is, protocol violations). Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | BF Spiromax | Symbicort Turbohaler
Number analyzed (Participants) | 289 | 284
L/min | 18.661 (2.631) | 21.740 (2.622)

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline up to Week 12
Population: The safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | BF Spiromax | Symbicort Turbohaler
Number analyzed (Participants) | 303 | 299
Participants | 117 | 106

4. Secondary Outcome: Number of Participants With Signs of Oral Candidiasis (Thrush)
Description: Examinations were performed by a qualified professional.
Time Frame: Baseline, Week 4, Week 8, Week 12
Population: The safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | BF Spiromax | Symbicort Turbohaler
Number analyzed (Participants) | 303 | 299
Participants
  Baseline | 0 | 0
  Week 4 | 1 | 0
  Week 8 | 1 | 2
  Week 12 | 2 | 3

5. Secondary Outcome: Number of Participants With Positive Swab of Oral Candidiasis (Thrush)
Description: Swab samples were collected by a qualified professional.
Time Frame: Baseline, Week 4, Week 8, Week 12
Population: The safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | BF Spiromax | Symbicort Turbohaler
Number analyzed (Participants) | 303 | 299
Participants
  Baseline | 1 | 0
  Week 4 | 0 | 0
  Week 8 | 0 | 0
  Week 12 | 1 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Description: The safety population included all randomized participants who received at least 1 dose of study medication.
Arm/Group | BF Spiromax | Symbicort Turbohaler
All-Cause Mortality (participants affected / at risk) | 0/303 | 0/299
Serious Adverse Events (participants affected / at risk) | 1/303 | 3/299
Other Adverse Events (participants affected / at risk) | 47/303 | 44/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BF Spiromax (N=303) | Symbicort Turbohaler (N=299)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BF Spiromax (N=303) | Symbicort Turbohaler (N=299)
Nasopharyngitis (Infections and infestations) | 31 (36) | 25 (27)
Headache (Nervous system disorders) | 18 (31) | 24 (57)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.